CLINICAL TRIAL: NCT01287832
Title: Vancomycin Versus Daptomycin for the Treatment of Methicillin-resistant Staphylococcus Aureus Bacteremia Due to Isolates With High Vancomycin Minimum Inhibitory Concentrations (MICs)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low patient enrollment
Sponsor: St. John Health System, Michigan (Other)
Collaborators: Henry Ford Health System (Other); Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Principal Investigator, Leonard B. Johnson, Division Chief, St. John Health System, Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ1210-01; IND 109,614 (Other: FDA)
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Bacteremia
Keywords: Methicillin-resistant; Staphylococcus aureus
MeSH Terms: conditions — Bacteremia; Staphylococcal Infections | interventions — Vancomycin; Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose vancomycin (Active Comparator): Vancomycin dosed to achieve a trough of 15-20 microgram/mL.
  Interventions: Drug: Vancomycin
- High-dose daptomycin (Experimental): Daptomycin dosed at 8 mg/kg/daily (every 48 hours in end-stage renal disease)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Vancomycin — Vancomycin dosed to achieve a trough of 15-20 microgram/mL.
  Arms: High dose vancomycin
Drug: Daptomycin
  Arms: High-dose daptomycin

SUMMARY:
There is an increased failure rate for the treatment of Staphylococcus Aureus Bacteremia (SAB) with traditional doses of vancomycin, the standard of care for patients with MRSA bacteremia over the last 40 years. This has been largely attributed to isolates with increased resistance to vancomycin (increased MIC). Daptomycin is an antibiotic that was approved several years ago for the treatment of SAB and is being increasingly used for MRSA bacteremia due to isolates with increased MIC. Increased doses have been recommended for both of these drugs in the treatment of this infection without a trial demonstrating their relative efficacy or safety at higher doses. This study will randomize patients with SAB due to MRSA with an increased MIC to determine the relative efficacy and safety of vancomycin and daptomycin used at higher than traditional doses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Signed informed consent
* All cases of suspected MRSA bacteremia as determined by a patient with at least one blood culture growing gram-positive cocci in clusters with a clinical syndrome consistent with true bacteremia including fever, hypothermia (temperature < 36.0º C), tachycardia (heart rate > 100 beats/minute), hypotension (systolic blood pressure < 90 mm Hg) or other clinical features of sepsis.
* All cases of right-sided native valve endocarditis due to MRSA
* Patients who are diagnosed with left-sided native valve endocarditis after randomization will be continued in the study
* Patients with MRSA bacteremia associated with infected foreign bodies, including vascular prostheses, orthopedic prostheses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Vancomycin: Vancomycin dosed to achieve a trough of 15-20 microgram/mL vs. daptomycin dosed at 8 mg/kg/daily (every 48 hours in end-stage renal disease)
Period: Overall Study
Arm/Group | High Dose Vancomycin | High-dose Daptomycin
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Dose Vancomycin; High-dose Daptomycin: Vancomycin vs. daptomycin: Vancomycin dosed to achieve a trough of 15-20 microgram/mL vs. daptomycin dosed at 8 mg/kg/daily (every 48 hours in end-stage renal disease)
- Total: Total of all reporting groups
Arm/Group | High Dose Vancomycin | High-dose Daptomycin | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (22.6) | 68.2 (10.2) | 64.7 (17.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Success at Test of Cure Visit.
Description: Clinical success is the absence of treatment failures. Treatment failures will include death, clinical failure, microbiologic failure, or an adverse event requiring a change in therapy or discontinuation in therapy.
Time Frame: 30-42 days post-treatment
Measure: Number; unit: participants
Arm/Group | High Dose Vancomycin | High-dose Daptomycin
Number analyzed (Participants) | 6 | 5
participants | 4 | 3

2. Secondary Outcome: Adverse Event Rate in Each Arm, Including the Nephrotoxicity and Skeletal Muscle Toxicity
Time Frame: 30-42 days post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Dose Vancomycin | High-dose Daptomycin
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vancomycin (N=6) | High-dose Daptomycin (N=5)
Nephrotoxicity (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Vancomycin (N=6) | High-dose Daptomycin (N=5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes